CLINICAL TRIAL: NCT06473623
Title: Non-invasive Auricular Fiber Vagus Nerve Stimulation (afVNS) for Treatment of Autism Spectrum Disorder: An Open-Label Trial
Brief Title: Non-invasive Auricular Fiber Vagus Nerve Stimulation (afVNS) for Treatment of Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuropix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 01A
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Receiving intervention of the non-invasive neurostimulation device.
  Interventions: Device: vagus nerve stimulation

INTERVENTIONS:
Device: vagus nerve stimulation — Non-invasive Auricular Fiber Vagus Nerve Stimulation (afVNS)

SUMMARY:
Non-invasive vagus nerve stimulation for the symptomatic improvements in Autism Spectrum Disorder

DETAILED DESCRIPTION:
A single arm open-label study in Autism Spectrum Disorder (ASD) for evaluating treatment effects of non-invasive VNS, specifically auricular fiber vagal nerve stimulation (afVNS). A total of 20 patients diagnosed with ASD will be recruited to evaluate the feasibility of home healthcare application of afVNS and for assessment of short-term treatment effects on symptoms and comorbidities. ASD patients will receive 1 x hour per day afVNS treatment over 14 days with a fixed neuromodulation protocol. The primary outcome measure is feasibility assessed from completion success and neurostimulation tolerance. Secondary outcome measures include changes in scores pre- and post- afVNS treatment for Clinician Global Clinical Impression (CGI-I), Clinician Global Impression Severity (CGI-S), Children's Anxiety Sensitivity Index (CASI-R), Parent-Rated Anxiety Scale for ASD (PRAS-ASD), Autistic Behavior Checklist (ABC), Cleveland Adolescent Sleep Questionnaire (CASQ), verbal fluency and biomarker measures in autonomic physiology.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age: between 7 and 26 years
* Participants and parent/ guardian must have proficiency in English
* Diagnosis of ASD as defined by ADOS-2 or DSM-5 criteria

Exclusion Criteria:

* Severe psychiatric disorders (e.g. bipolar, major depressive disorder)
* Severe neurological disorders (e.g. stroke, epilepsy)
* Bradyarrhythmia
* History of head trauma (surgery or tumor)
* Active medical implants (cochlear, VNS or pacemakers)
* Cerebral shunts
* Auricular skin disease that compromises placement of electrodes
* Pregnancy

Ages: 7 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility for completed treatments and stimulation intensity tolerance | 2 weeks
  Completion success and neurostimulation tolerance

SECONDARY OUTCOMES:
Clinician Global Clinical Impression (CGI-I) | 2 weeks
  For core social impairment and overall level of cognitive, adaptive and social functioning
Clinician Global Impression Severity (CGI-S) | 2 weeks
  For assessment of anxiety, gastrointestinal symptoms and social interactions and overall ASD
Parent-Rated Anxiety Scale for ASD (PRAS-ASD) | 2 weeks
  For anxiety assessment consisting of 25 questions related to anxiety ranging from 0 (none) to 3 (severe)
Autistic Behavior Checklist (ABC) scores | 2 weeks
  For measurements of 5 behavioral domains including irritability, social withdrawal, stereotypy, hyperactivity and inappropriate speech

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Ko, PhD, Principal Investigator — Neuropix
Locations (1):
- Hong Kong Science Park, Tai Po, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jin Y, Kong J. Transcutaneous Vagus Nerve Stimulation: A Promising Method for Treatment of Autism Spectrum Disorders. Front Neurosci. 2017 Jan 20;10:609. doi: 10.3389/fnins.2016.00609. eCollection 2016. PMID 28163670
- [Background] Black B, Hunter S, Cottrell H, Dar R, Takahashi N, Ferguson BJ, Valter Y, Porges E, Datta A, Beversdorf DQ. Remotely supervised at-home delivery of taVNS for autism spectrum disorder: feasibility and initial efficacy. Front Psychiatry. 2023 Sep 28;14:1238328. doi: 10.3389/fpsyt.2023.1238328. eCollection 2023. PMID 37840787
- [Background] Molero-Chamizo A, Nitsche MA, Bolz A, Andujar Barroso RT, Alameda Bailen JR, Garcia Palomeque JC, Rivera-Urbina GN. Non-Invasive Transcutaneous Vagus Nerve Stimulation for the Treatment of Fibromyalgia Symptoms: A Study Protocol. Brain Sci. 2022 Jan 12;12(1):95. doi: 10.3390/brainsci12010095. PMID 35053839

DOCUMENTS (2):
  • Study Protocol (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT06473623/Prot_000.pdf
  • Statistical Analysis Plan (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT06473623/SAP_001.pdf